CLINICAL TRIAL: NCT04168385
Title: MRX-800: A Long-Term Safety Study of Maralixibat, an Apical Sodium Dependent Bile Acid Transporter Inhibitor (ASBTi), in the Treatment of Cholestatic Liver Disease in Subjects Who Previously Participated in a Maralixibat Study
Brief Title: MRX-800: A Long-Term Safety Study of Maralixibat in the Treatment of Cholestatic Liver Disease in Subjects Who Previously Participated in a Maralixibat Study
Acronym: MERGE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mirum Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRX-800
Record Dates: First submitted 2019-10-01; First posted 2019-11-19 (Actual); Results first posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Cholestatic Liver Disease
Keywords: PFIC; ALGS; Maralixibat; Bile Duct Diseases; Liver Diseases; Biliary Tract Diseases; Digestive System Diseases; Pediatric
MeSH Terms: conditions — Bile Duct Diseases; Liver Diseases; Biliary Tract Diseases; Digestive System Diseases | interventions — maralixibat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Maralixibat (Experimental): Participants will all receive Maralixibat oral solution
  Interventions: Drug: Maralixibat

INTERVENTIONS:
Drug: Maralixibat — Maralixibat chloride oral solution orally twice daily (up to 1200* mcg/kg/day), and according to indication.
  *equivalent to 1140 mcg/kg/day maralixibat
  Other Names: Formerly LUM001 and SHP625

SUMMARY:
Evaluate the long-term safety of maralixibat (MRX) in subjects with cholestatic liver disease including, but not limited to, Alagille Syndrome (ALGS), Progressive Familial Intrahepatic Cholestasis (PFIC) and Biliary Atresia.

DETAILED DESCRIPTION:
This is a multicenter, open-label study of maralixibat in subjects diagnosed with cholestatic liver disease (including, but not limited to ALGS, PFIC or Biliary Atresia) who have previously participated in a maralixibat clinical study. All subjects received maralixibat in the previous studies and will continues to receive maralixibat in this study.

ELIGIBILITY:
Inclusion Criteria Subjects will need to meet all criteria below to be considered eligible for the study.

1. Provide informed consent and assent (as applicable) per the Institutional Review Board/Ethics Committee (IRB/EC).
2. Previously participated in a maralixibat study and with approval of the Medical Monitor. Previous participation is defined as:

   * Having completed the EOT Visit, for subjects coming from the maralixibat Phase 2 studies.
   * Having completed the entire duration of the study (i.e., core and extension, if applicable), for subjects coming from the maralixibat Phase 3 studies.
3. At least 1 year of age
4. Males, and females of non-childbearing potential. Males and non-pregnant, non-lactating females of childbearing potential who are sexually active must agree to use acceptable contraception during the study and 30 days following the last dose of the study medication. Females of childbearing potential must have a negative pregnancy test.
5. Caregivers (and/or age appropriate subjects) must have access to email or phone for scheduled remote visits if applicable.
6. Subject and caregiver willingness to comply with all study visits and requirements.

Exclusion Criteria

A subject will be excluded from the study if any of the following exclusion criteria are met:

1. Experienced an AE or SAE related to maralixibat during the lead-in protocol that led to permanent discontinuation of the subject from maralixibat.
2. Any conditions or abnormalities (including laboratory abnormalities) which, in the opinion of the Investigator or Medical Monitor may compromise the safety of the subject or interfere with the subject participating in or completing the study.
3. History of non-adherence to medical regimens, unreliability, medical condition, mental instability or cognitive impairment that, in the opinion of the Investigator or Sponsor medical monitor, could compromise the validity of informed consent, compromise the safety of the subject, or lead to non-adherence with the study protocol or inability to conduct the study procedures.

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2024-09-04 (Actual); Study Completion 2024-09-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (6):
  - Children'S Hospital Los Angeles, Los Angeles, California
  - Riley Hospital For Children, Indianapolis, Indiana
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Baylor College of Medicine/Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Australia (2):
  - Children's Hospital Westmead, Westmead, New South Wales
  - The Royal Children'S Hospital Melbourne, Parkville, Victoria
- Cliniques Universitaires Saint-Luc, Brussels, Belgium
- Hospital for Sick Children, Toronto, Canada
- France (2):
  - Hopital Necker-Enfants Malades, Paris
  - Hopital Kremlin Bicetre, Paris
- The Children's Memorial Health Institute, Warsaw, Poland
- Hospital Universitario La Paz- Hospital Materno Infantil, Madrid, Spain
- United Kingdom (3):
  - Birmingham Children's Hospital, Birmingham
  - Leeds Teaching Hospital NHS Trust, Leeds
  - Paediatric Liver Center, Kings College Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Genetics Home Reference - PFIC — https://ghr.nlm.nih.gov/condition/progressive-familial-intrahepatic-cholestasis
- See also: Genetics Home Reference - Alagille syndrome — https://ghr.nlm.nih.gov/condition/alagille-syndrome
- See also: US FDA Resources — https://clinicaltrials.gov/ct2/info/fdalinks
- See also: Mirum Pharmaceuticals homepage — https://mirumpharma.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 52 participants were enrolled at 17 sites across 8 countries (Australia, Belgium, Canada, France, Poland, Spain, United Kingdom and United States). Participants were previously on maralixibat for an average of 4 years before entering this study.
Pre-assignment Details: The screening period starts when informed consent (by the legally authorized representative) is signed.The duration of the screening period is up to 4 weeks, during which all procedures listed for the screening visit in the schedule of assessment must be completed. A total of 43 subjects completed the study and a total of 9 discontinued early.
Groups:
- Maralixibat: ALGS: Participants will all receive Maralixibat oral solution
  Maralixibat chloride oral solution orally twice daily Up to 1.2* mg/kg/day), and according to indication.
  *equivalent to 1.14 mg/kg/day maralixibat. Doses reported here are in maralixibat chloride.
  Participants with ALGS received maralixibat doses in the range of 0.15 mg/kg QD to 0.45 mg/kg BID.
- Maralixibat: PFIC: Participants will all receive Maralixibat oral solution
  Maralixibat chloride oral solution orally twice daily Up to 1.2* mg/kg/day), and according to indication.
  *equivalent to 1.14 mg/kg/day maralixibat. Doses reported here are in maralixibat chloride.
  Participants with PFIC received maralixibat doses in the range of 0.3 mg/kg QD to 0.6 mg/kg BID.
Period: Overall Study
Arm/Group | Maralixibat: ALGS | Maralixibat: PFIC
Started | 40 | 12
Completed | 33 | 10
Not Completed | 7 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 2 | 1
Not completed — Liver transplant | 3 | 1
Not completed — Listed for liver transplant | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Maralixibat: ALGS | Maralixibat: PFIC | Total
Number analyzed (Participants) | 40 | 12 | 52
Age, Customized [Count of Participants; unit: Participants]
  Age Categorical: 5 to 8 years | 8 | 4 | 12
  Age Categorical: 9 to 12 years | 18 | 7 | 25
  Age Categorical: 13 to 18 years | 9 | 1 | 10
  Age Categorical: > 18 years | 5 | 0 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 7 | 26
  Male | 21 | 5 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 6
  Not Hispanic or Latino | 21 | 11 | 32
  Unknown or Not Reported | 14 | 0 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 22 | 10 | 32
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 15 | 0 | 15
Region of Enrollment [Number; unit: participants]
  Canada | 2 | 0 | 2
  Belgium | 2 | 0 | 2
  United States | 18 | 8 | 26
  Poland | 1 | 1 | 2
  United Kingdom | 8 | 3 | 11
  Australia | 4 | 0 | 4
  France | 4 | 0 | 4
  Spain | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-Emergent Adverse Events
Description: TEAE = Treatment-emergent Adverse Event; AESI = Adverse Event of Special Interest..
Time Frame: From informed consent through approximately 4.5 years, including 30 days after last dose.
Population: Includes all participants with Alagille Syndrome (ALGS) or Progressive Familial Intrahepatic Cholestasis (PFIC) who received at least one dose of maralixibat.
Measure: Count of Participants; unit: Participants
Arm/Group | Maralixibat: ALGS | Maralixibat: PFIC
Number analyzed (Participants) | 40 | 12
Participants
  At least one TEAE | 36 | 12
  TEAE ≥ 3 | 9 | 4
  Serious TEAE | 10 | 3
  Serious Treatment-Related Adverse Event | 0 | 0
  Serious Treatment-Related TEAE | 0 | 0
  TEAE Leading to Discontinuation of Study Drug | 3 | 1
  TEAE Leading to Death | 1 | 0
  Treatment-emergent AESI | 0 | 1

2. Secondary Outcome: Long-Term Effect on Pruritus
Description: Change from Baseline in Pruritus Severity assessed using the Clinician Scratch Score (CSS), a 5-point scale where 0 indicates no evidence of scratching and 4 indicates cutaneous mutilation with bleeding, hemorrhage, and scarring.
Time Frame: From Baseline through Week 160, including Change from Baseline values.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Maralixibat: ALGS | Maralixibat: PFIC
Number analyzed (Participants) | 40 | 12
score on a scale | -0.4 (0.89) | -0.3 (1.12)

3. Secondary Outcome: Long-Term Effect on Serum Bile Acid Levels
Time Frame: From Baseline through Week 160, including Change from Baseline values.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µmol/L
Groups:
- Maralixibat: ALGS: Maralixibat chloride oral solution orally twice daily Up to 1.2* mg/kg/day), and according to indication.
  *equivalent to 1.14 mg/kg/day maralixibat. Doses reported here are in maralixibat chloride.
  Participants with ALGS received maralixibat doses in the range of 0.15 mg/kg QD to 0.45 mg/kg BID
- Maralixibat: PFIC: Maralixibat chloride oral solution orally twice daily Up to 1.2* mg/kg/day), and according to indication.
  *equivalent to 1.14 mg/kg/day maralixibat. Doses reported here are in maralixibat chloride.
  Participants with PFIC received maralixibat doses in the range of 0.3 mg/kg QD to 0.6 mg/kg BID
- Maralixibat: Overall: Combined results of ALGS and PFIC Groups
Arm/Group | Maralixibat: ALGS | Maralixibat: PFIC | Maralixibat: Overall
Number analyzed (Participants) | 40 | 12 | 52
µmol/L | -15.948 (31.4239) | -82.647 (136.4354) | -59.994 (111.0334)

ADVERSE EVENTS:
Time Frame: The timeframe for reporting adverse events was from informed consent through approximately 4.5 years, including 30 days after last dose.
Arm/Group | Maralixibat: ALGS | Maralixibat: PFIC
All-Cause Mortality (participants affected / at risk) | 1/40 | 0/12
Serious Adverse Events (participants affected / at risk) | 10/40 | 3/12
Other Adverse Events (participants affected / at risk) | 36/40 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maralixibat: ALGS (N=40) | Maralixibat: PFIC (N=12)
Alagille syndrome (Congenital, familial and genetic disorders) | 2 (2) | 0 (0)
Arteriovenous malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Coarctation of the aorta (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Abdominal mass (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Condition aggravated (General disorders) | 0 (0) | 1 (2)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Lung abscess (Infections and infestations) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nodular lymphocyte predominant Hodgkin lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Fibrinous bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hepatopulmonary syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maralixibat: ALGS (N=40) | Maralixibat: PFIC (N=12)
Splenomegaly (Blood and lymphatic system disorders) | 3 (4) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 2 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 6 (10) | 3 (7)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2)
Dental caries (Gastrointestinal disorders) | 1 (1) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 4 (7)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (6) | 0 (0)
Pancreatic failure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 2 (2) | 3 (4)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Fatigue (General disorders) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 2 (3) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 7 (10) | 2 (4)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic mass (Hepatobiliary disorders) | 5 (5) | 0 (0)
Liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Allergy to arthropod sting (Immune system disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 4 (6) | 0 (0)
Corona virus infection (Infections and infestations) | 9 (10) | 9 (14)
Ear infection (Infections and infestations) | 2 (3) | 2 (2)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 1 (1)
Impetigo (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (2) | 1 (1)
Lung abscess (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 7 (16) | 4 (6)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 2 (4) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 2 (3)
Upper respiratory tract infection (Infections and infestations) | 4 (5) | 5 (8)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (2) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Oral contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Stress fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 3 (5) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Anti-transglutaminase antibody increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Bilirubin conjugated increased (Investigations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 2 (4)
Blood phosphorus decreased (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 2 (6)
Spleen scan abnormal (Investigations) | 0 (0) | 1 (1)
Ultrasound liver abnormal (Investigations) | 2 (2) | 1 (1)
Vitamin A decreased (Investigations) | 2 (2) | 0 (0)
Vitamin D decreased (Investigations) | 2 (3) | 1 (1)
Weight decreased (Investigations) | 2 (2) | 0 (0)
Vitamin A deficiency (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Vitamin E deficiency (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Epiphyses delayed fusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Growing pains (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (5) | 3 (4)
Head discomfort (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 3 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (11) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Milia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-11-16): https://cdn.clinicaltrials.gov/large-docs/85/NCT04168385/Prot_003.pdf
  • Statistical Analysis Plan (2024-09-06): https://cdn.clinicaltrials.gov/large-docs/85/NCT04168385/SAP_004.pdf